CLINICAL TRIAL: NCT03812692
Title: Validation of a Simplified MATRx Plus Theragnostic Sleep Study
Brief Title: Validation of a Simplified MATRx Plus
Status: Completed | Type: Observational
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: ZCP201901
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral appliance therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- MATRx plus test: All participants will complete the MATRx plus test unattended in the home. Not all participants will be predicted responders to oral appliance therapy; both predicted responders and non-responders will undergo an outcome home sleep apnea test with a custom oral appliance in place to validate the prediction made by the test. Twenty participants will also complete an in-lab sleep study prior to the home study.
  Interventions: Device: MATRx plus

INTERVENTIONS:
Device: MATRx plus — The MATRx plus device is a feedback-controlled mandibular positioner that uses data collected during sleep to control movement of the mandible in real-time using a mandibular positioner. The test provides a prediction of the individual's response to oral appliance therapy; i.e., if the individual can treat his or her obstructive sleep apnea using a mandibular advancing oral appliance. For individuals predicted to respond to the therapy, the test also provides a mandibular position at which the appliance will be effective.

SUMMARY:
Sleep apnea (OSA) is a condition in which the air passage in the throat closes or partly closes during sleep and repeatedly interrupts breathing. The standard treatment for sleep apnea is continuous positive airway pressure (CPAP), but it is not suitable for all patients. Another treatment is to use an oral appliance in your mouth when you sleep. The appliance covers the upper and lower teeth and acts to pull the lower jaw forward, opening the throat passage and allowing normal breathing.

Oral appliance therapy does not treat sleep apnea effectively in everyone. In order to identify the people in whom oral appliance therapy will work, Zephyr Sleep Technologies has invented a feedback-controlled device that tests various positions of the lower jaw. This commercially available device, known as MATRx plus, is a Health Canada approved and FDA cleared motorized dental positioner that can be used in an overnight sleep study performed in the home. Temporary dental impression trays cover your upper and lower teeth. These are attached to a small motor that slowly and gently pulls your lower jaw forward under the control of a computer in response to real-time breathing events. The commercial MATRx plus device uses measures of airflow from a nasal cannula and blood oxygen saturation from a pulse oximeter to guide the movement of the lower jaw during the test. Though the test is accurate, the equipment can be somewhat cumbersome to apply. The purpose of the study is to validate a simplified version of the test that requires fewer sensors and sleep time.

DETAILED DESCRIPTION:
Sleep apnea (OSA) is a condition in which the air passage in the throat closes or partly closes during sleep and repeatedly interrupts breathing. The standard treatment for sleep apnea is continuous positive airway pressure (CPAP), but it is not suitable for all patients. Another treatment is to use an oral appliance in your mouth when you sleep. The appliance covers the upper and lower teeth and acts to pull the lower jaw forward, opening the throat passage and allowing normal breathing.

Oral appliance therapy does not treat sleep apnea effectively in everyone. In order to identify the people in whom oral appliance therapy will work, Zephyr Sleep Technologies has invented a feedback-controlled device that tests various positions of the lower jaw. This commercially available device, known as MATRx plus, is a Health Canada approved and FDA cleared motorized dental positioner that can be used in an overnight sleep study performed in the home. Temporary dental impression trays cover your upper and lower teeth. These are attached to a small motor that slowly and gently pulls your lower jaw forward under the control of a computer in response to real-time breathing events. The commercial MATRx plus device uses measures of airflow from a nasal cannula and blood oxygen saturation from a pulse oximeter to guide the movement of the lower jaw during the test. Though the test is accurate, the equipment can be somewhat cumbersome to apply. The purpose of the study is to validate a simplified version of the test that requires fewer sensors and sleep time.

We have previously carried out three research studies leading to the development of the feedback-controlled mandibular positioner. These studies, two of which used early prototypes of the device and one that used the commercial MATRx plus device, showed that the feedback-control software used was very accurate and was able to identify successful candidates in a home setting.

No serious or permanent problems or risks were identified in any of the previous research studies. Participants reported minor tooth and gum discomfort on the morning following the test and other minor issues including dry mouth, excessive saliva, and being unable to sleep. The previous studies have established the safety and efficacy of the device using a device prototype. The purpose of the present study is to determine if the efficacy of the device is maintained when fewer sensors are used and the requirement for sleep time is reduced.

The study will collect data over one night in a sleep laboratory and a series of nights in the home. Following the study, you will be told if you are a suitable candidate for oral appliance therapy. If you do not already have a custom oral appliance, one will be provided to you. During the study, the Principal Investigator and study dentist will be blinded to the results of your tests. In the event of an emergency, the Principal Investigator can be unblinded to your test results.

Up to 46 individuals will be recruited for this study. Study participants will need to attend visits at multiple centres located in Calgary, Alberta.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 21 and 80 years
2. Obstructive sleep apnea (ODI > 10 h-1)
3. Body mass index < 45 kg/m2
4. Neck circumference < 50 cm
5. Absence of severe oxyhemoglobin desaturation during sleep, indicated by a mean value of oxyhemoglobin saturation (SaO2) > 87%
6. Mandibular range of motion > 5 mm
7. Adequate dentition (10 upper and 10 lower teeth)
8. Ability to understand and provide informed consent
9. Ability and willingness to meet the required schedule

Exclusion Criteria:

1. Inability to breathe comfortably through the nose
2. Central Sleep Apnea (> 50% of apneas are central)
3. Anticipated change in medical therapy that could alter the severity of OSA during the protocol
4. Anticipated change in body weight (5% or more) during the protocol
5. Symptomatic, non-respiratory sleep disorder, e.g., restless leg syndrome or chronic insomnia
6. Severe respiratory disorder(s) other than sleep disordered breathing
7. Loose teeth, faulty restorations, or advanced periodontal disease
8. Participation in other studies that could interfere with study protocol
9. Pregnant or nursing
10. Heart failure
11. Cerebral vascular incident within the last 12 months
12. Use of pacemaker or other life supporting device
13. Regular use of CPAP or oral appliance therapy within 5 days of the PSG or HSAT (individuals on therapy wishing to participate may opt to cease therapy for the 5 nights prior to each test)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be representative of the general population of individuals with obstructive sleep apnea in North America.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Oxygen desaturation index | 6 weeks
  With the oral appliance in place, participants will complete a 2-night home sleep apnea test with a Level III sleep recorder. The participant's oxygen desaturation index with the appliance will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Zephyr Sleep Technologies, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mosca EV, Grosse J, Remmers JE. Oral appliance therapy is highly efficacious at reducing sleep apnea-specific hypoxic burden, a metric predictive of cardiovascular morbidity and mortality. J Clin Sleep Med. 2025 Jul 1;21(7):1185-1190. doi: 10.5664/jcsm.11622. PMID 40123555